CLINICAL TRIAL: NCT00883610
Title: Modulation of QT Interval by Rapid Atrial Pacing in Patients With Dual Chamber Pacemakers
Brief Title: Effects Rapid Atrial Pacing Has on the Electrocardiogram (ECG) in Patients With Dual Chamber Pacemakers
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Dawood Darbar, Associate Professor of Medicine and Clinical Pharmacology, Vanderbilt University
Other Study IDs: 070070
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Prolonged QT Interval
Keywords: QT Interval; Dual Chamber Pacemaker; Atrial Fibrillation
MeSH Terms: conditions — Long QT Syndrome; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to learn what effect rapid atrial pacing (in patients with dual chamber pacemakers) will have on the electrocardiogram including the QT Interval. The investigators are also interested in the differences caused by genes.

DETAILED DESCRIPTION:
This study requires a total of two study days as well as two follow up visits. During study day one, baseline blood will be drawn, a baseline electrocardiogram will be performed, and continuous QT Interval monitoring will be performed. The pacemaker rate will be increased to 90bpm at different time intervals and additional blood will be drawn to measure the effects of these rates changes.

On study day two, baseline blood will be drawn, a urine specimen will be obtained, an electrocardiogram will be performed, and continuous QT Interval monitoring will be performed. Following the acquisition of this information, the pacemaker rate will be decreased to 80bpm. We will obtain blood specimens, a urine specimen and an electrocardiogram at 30 minutes post rate change and again at 60 minutes post rate change.

Two days following the rate decrease to 80bpm, the patient will return to clinic to have their rate decreased to 70bpm. In two more days, the patient will return for a final rate change to 60bpm.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 21 years old
* Must have a dual chamber pacemaker implanted more than three months ago
* Must be followed by the Vanderbilt University Medical Center's Arrhythmia Device Clinic
* The indication for the pacemaker must not be related to coronary artery disease (CAD) or congestive heart failure (CHF)

Exclusion Criteria:

* Cannot be pacemaker dependent
* History of ventricular arrhythmias and/or implantable defibrillators (ICDs)
* History of paroxysmal, persistent, or permanent atrial fibrillation (AF)
* Congenital long QT syndrome
* History of coronary artery disease
* History of, or currently receiving, treatment for congestive heart failure
* Unable to tolerate dual-chamber pacing (DDD) at 90 bpm due to palpitations, chest pain, shortness of breath, lightheadedness, dizziness, or presyncope
* Pregnant women
* Any patient without specific documentation of an echocardiogram negative for CHF (systolic or diastolic dysfunction)within five years prior to study enrollment
* Any patient without specific documentation of an objective diagnostic test to rule out CAD within five years prior to study enrollment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiology Clinic
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Determine the effect of abrupt changes in atrial rate on QT intervals | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Dawood Darbar, M.D., Ph.D., F.A.C.C., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States